CLINICAL TRIAL: NCT01591395
Title: Prospective Randomized Trial Comparing the Short-term and Long-term Outcomes of Three-port and Single-port TEP Repair in Adults
Brief Title: Prospective Randomized Trial Comparing Three-port and Single-port TEP Repair in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Yao-Chou Tsai, Principle investigator, M.D., Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99-IRB-003-X
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; laparoscopy; laparoendoscopic single-site surgery
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiport TEP (Active Comparator): Adult inguinal hernia patients who randomized to receive multiport endoscopic TEP repair
  Interventions: Procedure: laparoscopic total extraperitoneal hernia repair (single port vs. multiport)
- LESS TEP (Active Comparator): Adult inguinal hernia patients who randomized to receive laparoendoscopic single-site TEP repair
  Interventions: Procedure: laparoscopic total extraperitoneal hernia repair (single port vs. multiport)

INTERVENTIONS:
Procedure: laparoscopic total extraperitoneal hernia repair (single port vs. multiport) — comparison of single port laparoscopic TEP and multiport laparoscopic TEP repair for adult inguinal hernia

SUMMARY:
Inguinal hernia is one of the most common surgical diseases. Over the past years, the safety and feasibility of laparoscopy was established and gaining popularity in recent few years. Laparoscopic inguinal hernia repair was associated with less post operative pain, a shorter recovery period, earlier return to normal daily activities and work, and better cosmetic results. The laparoscopic hernia repair usually require three working ports ranging from 5 to 10 mm. However, with each increasing laparoscopic ports usually associated with possible increasing morbidity and pain related to ports.

Efforts are continuing to further reduce the port related morbidities and improve the cosmetic outcomes of laparoscopic surgery, including reduction of the size and number of ports. This has led to the evolution of a novel surgical approach now collectively known as laparoendoscopic single site surgery. LESS has been performed for variable indications including extirpative and reconstructive urologic procedure via the transperitoneal approach. Early experience has demonstrated the feasibility as well as the safe and successful completion of these LESS procedures. Although these initial reports are promising, the clinical advantages of LESS procedures over conventional laparoscopic procedures have not been defined. Therefore, we conducted a single center, randomized trial to compare the safety and other outcomes after conventional laparoscopic and LESS inguinal hernia repair in adult patients.

DETAILED DESCRIPTION:
Inguinal hernia is one of the most common surgical diseases in adult. Tension free hernioplasty is regarded as gold standard of treatment in adult inguinal hernia. The reported incidence of hernia recurrence after tension free repair is less than 5 percent. Over the past years, the safety and feasibility of laparoscopy was established and gaining popularity in recent few years. With the advancing technology, laparoscopic approach has become the standard treatment for cholecystectomy and adrenalectomy. Laparoscopic procedures improved surgical precision through enhanced visualization, magnification and limited exposure, dissection. Laparoscopic inguinal hernia repair was associated with less postoperative pain, a shorter recovery period, earlier return to normal daily activities and work, and better cosmetic results. The laparoscopic hernia repair usually require three working ports ranging from 5 to 10 mm. However, with each increasing laparoscopic ports usually associated with possible increasing morbidity and pain related to ports.

Efforts are continuing to further reduce the port related morbidities and improve the cosmetic outcomes of laparoscopic surgery, including reduction of the size and number of ports. This has led to the evolution of a novel surgical approach now collectively known as laparoendoscopic single-site surgery. LESS has been performed for variable indications including extirpative and reconstructive urologic procedure via the transperitoneal approach. Early experience has demonstrated the feasibility as well as the safe and successful completion of these LESS procedures. Although these initial reports are promising, the clinical advantages of LESS procedures over conventional laparoscopic procedures have not been defined.

To date, LESS hernia repair had been rarely reported in the literature except in some case reports and one small series. Although these initial reports revealed that LESS hernia repair is safe and feasible in adult inguinal hernia, the definite clinical benefits of LESS hernia repair could not be identified in these small and short term reports. Thus, a prospective randomized trial comparing LESS and conventional multiport laparoscopic hernia repair with long-term follow up was mandatory to define the clinical advantages of LESS hernia repair. Therefore, we conducted a randomized trial to compare LESS total extraperitoneal hernia repair and conventional multiport TEP repair in adult inguinal hernia with inflammatory, gonadal responses, complication rate and recurrence rate and pain score, functional status and activity level.

Overall Goal

-To compare the surgical outcomes, patient center outcomes and surgery induced inflammatory , gonadal responses after LESS TEP and conventional multiport TEP hernia repair in adult.

Specific Aims

* Compare the surgery induced inflammatory responses after LESS TEP and conventional multiport TEP hernia repair with inflammatory markers by blood sampling before and after operation.
* Compare the surgery induced testicle changes in male adults after LESS TEP and conventional multiport TEP hernia repair with color Doppler ultrasonography to determine testicular volume and resistive index before surgery and 3 months postoperatively.
* Compare the postoperative pain score after LESS TEP and conventional multiport TEP hernia repair with Visual analog pain score.
* Compare the postoperative activity level after LESS TEP and conventional multiport TEP hernia repair with modified Medical Outcome Study.
* Compare the clinical results and complication rates after LESS TEP and conventional multiport TEP hernia repair by clinic follow up.
* Compare the longterm functional outcomes 6 months after LESS TEP and conventional multiport TEP hernia repair with follow up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* primary or recurrent inguinal hernia

Exclusion Criteria:

* previous major lower abdominal surgery, patient refusal of randomization, or unable to accept general anesthesia

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain score | 7 days post-operatively
  The pain score was recorded by a blinded observer at the time points of 2 hours post-op, 24 hours post-op and 7 days post-op with a Visual analoge pain scale (0-10 scale)

SECONDARY OUTCOMES:
modified Medical Outcome Study (MOS) | Post -op 6 months
  The post-op convalescence was evaluated by a Modified medical outcome study with item 3-12. The time points being evaluated are at 1 day after operation, 7 days after operation and 6 months after operation.
systemic stress response to surgery | post-operative 1 day
  Compare the surgery induced inflammatory responses after LESS TEP and conventional multiport TEP hernia repair with inflammatory markers (IL-6, CRP and neutrophil counts) by blood sampling before and after operation
Testicular volume | 3 months post-operatively
  Compare the surgery induced testicle changes in male adults after LESS TEP and conventional multiport TEP hernia repair with color Doppler ultrasonography to determine testicular volume and resistive index (RI) before surgery and 3 months postoperatively.
intervention related complication | 6 months post-operatively
  wound infection, ecchymosis of skin, bleeding complication, seroma formation, chronic wound pain..etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Chou Tsai, Principal Investigator — 289 Jianguo Road, Xindian city, Taipei, Taiwan
Locations (1):
- Buddhist Tzu Chi General Hospital, Taipei branch, Taipei, Taiwan, Taiwan